Statistical Analysis Plan: ACE-ST-209

Version 1.0 dated:07 April 2018

Protocol Number: ACE-ST-209

Protocol Title: A Phase 1b/2, Multicenter, Open-label Study of ACP-196

in Subjects with Recurrent Glioblastoma Multiforme (GBM)

Version: 1.0

Version date: 07 April 2018

The undersigned have reviewed this plan and find it to be consistent with the requirements of the protocol as it applies to their respective areas



#### **CONFIDENTIAL**

This document (and all copies thereof) is the property of Acerta Pharma and contains valuable trade secrets and confidential information, including proprietary technical and business information. By accepting this document, you agree that the Confidential Information contained herein will not be disclosed to others without prior written authorization from Acerta Pharma and shall only be used for the purposes intended by the document.

Product: Acalabrutinib Statistical Analysis Plan: ACE-ST-209 Version 1.0 dated:07 April 2018

# Statistical Analysis Plan

A Phase 1b/2, Multicenter, Open-label Study of ACP-196 in Subjects with Recurrent Glioblastoma Multiforme (GBM)

**Protocol Number ACE-ST-209** 

Version: Date: 1.0 07 April 2018


**Study Statistician:** 

Acerta Pharma Confidential

# **TABLE OF CONTENTS**

| Tabl | Table of Contents | |
|---|---|---|
| Tabl | Table of Abbreviations4 | |
| 1 | INTRODUCTION | 6 |
| 2 | OBJECTIVES | 6<br>6 |
| 3 | STUDY OVERVIEW 3.1 Study Design 3.2 Sample Size. | 6 |
| 4 | STUDY ENDPOINTS | .8<br>.9 |
| 5 | HYPOTHESES AND MULTIPLICITY | .9 |
| 6 | ANALYSIS SETS | .9 |
| 7 | SUBGROUP ANALYSIS | .9 |
| 8 | FINAL ANALYSIS AND CLINICAL STUDY REPORT | .9 |
| 9 | MISSING VALUES9 | |
| 10 | STATISTICAL METHODS OF ANALYSIS 10.1 General Principles 10.2 Subject Accountability 10.3 Important Protocol Deviations 10.4 Demographic and Baseline Characteristics 10.5 Treatment and Medications 10.5.1 Prior Anticancer Therapies 10.5.2 Concomitant Medications 10.5.3 Exposure to Investigational Product 10.6 Safety Analyses 10.6.1 Adverse Events | 10<br>10<br>10<br>10<br>11<br>11<br>11 |
| | 10.6.2 Events of Clinical Interest | |

| | 10.6.3 | Laboratory Test Results | 12 |
|---|---|---|---|
| | 10.6.4 | Vital Signs | 12 |
| | 10.6.5 | ECOG Performance Status | 12 |
| | 10.7 Efficacy | y Analyses | 12 |
| | 10.7.1 | Best Overall Response, Disease Control Rate and Overall Response Rate per RANO criteria | 13 |
| | 10.7.2 | Duration of Response per RANO criteria | 13 |
| | 10.7.3 | Progression-free Survival Per RANO criteria | 13 |
| | 10.7.4 | Overall Survival | 14 |
| | 10.7.5 | Pharmacokinetic, Pharmacodynamic and Biomarker Analyses | 15 |
| 11 | LITERATURI | E CITATIONS / REFERENCES | 16 |
| 12 | APPENDICE | s | 17 |
| | 12.1 Definitions | | |
| | 12.2 Imputat | ion rules for partial or missing dates | 18 |
| | 12.3 PFS ev | ents and censoring rules | 19 |
| | 12.4 Overall | survival censoring rules | 20 |
| | 12.5.1 Eve | nts of Clinical Interest | 21 |
| | 12.5.2 Maid | or Hemorrhage | 22 |

Statistical Analysis Plan: ACE-ST-209 Version 1.0 dated:07 April 2018

#### **TABLE OF ABBREVIATIONS**

ACP-196 Acalabrutinib (acalabrutinib = ACP-196)

AE adverse event

BID twice per day (dosing)
BMI body mass index

CCNU Iomustine

CI confidence interval

CR complete response (remission)

CRF case report form
CSR clinical study report

CTCAE Common Terminology Criteria for Adverse Events

DOR duration of response

ECOG Eastern Cooperative Oncology Group

ECI Events of Clinical Interest

EIAEDs enzyme-inducing antiepileptic drugs

FACT-Br Functional Assessment of Cancer Therapy – Brain

FDA Food and Drug Administration

GBM Glioblastoma Multiform
ICF Informed Consent Form
IPD Important Protocol Deviation

K-M Kaplan-Meier

MDSCs myeloid-derived suppressor cells

MedDRA Medical Dictionary for Regulatory Activities

mmHG millimeter of mercury

NCI National Cancer Institute

ORR overall response rate

OS overall survival

PD pharmacodynamic, pharmacodynamics, or progressive disease

PFS progression-free survival

PFS-4 4-month progression-free survival
PFS-6 6-month progression-free survival
PK pharmacokinetic or pharmacokinetics

PO orally

PR partial response (remission)
PRO patient-reported outcome

PT preferred terms

QD once per day (dosing)

RANO Response Assessment in Neuro-oncology (criteria)

RCI Reliable Change Index (methodology)

SAC Scientific Advisory Committee

SAE serious adverse event SAP statistical analysis plan

SD stable disease

Acerta Pharma 

Statistical Analysis Plan: ACE-ST-209


SI International System of Units

SMQ Standardized MedDRA Queries

SOC system organ class

SRC Safety Review Committee

TEAEs treatment emergent adverse events

TESAEs treatment-emergent serious adverse events

WHO World Health Organization

WHODRUG World Health Organization Drug Dictionary

Statistical Analysis Plan: ACE-ST-209


#### 1 INTRODUCTION

The purpose of this statistical analysis plan (SAP) is to provide details of the statistical analyses that have been outlined within the protocol Amendment 2.0, 21 March 2017 for ACE-ST-209 (Glioblastoma multiforme, GBM). The scope of this plan includes the final analysis that are planned and will be executed by the Biometrics department or designee. Any changes to the methods described in the final SAP will be documented in the clinical study report (CSR).

#### 2 OBJECTIVES

### 2.1 Primary Objectives

- To characterize the safety profile of acalabrutinib monotherapy in subjects with recurrent GBM
- To evaluate the efficacy of acalabrutinib monotherapy in subjects with recurrent GBM based on overall response rate (ORR) per the Response Assessment in Neuro-oncology (RANO) criteria

# 2.2 Secondary Objectives

- To evaluate the efficacy of acalabrutinib monotherapy based on duration of response (DOR) per RANO criteria
- To evaluate the efficacy of acalabrutinib monotherapy based on progressionfree survival (PFS) per RANO criteria
- To evaluate the efficacy of acalabrutinib monotherapy based on 6-month PFS (PFS-6) rate per RANO criteria
- To evaluate the efficacy of acalabrutinib monotherapy based on overall survival (OS)

# 2.3 Exploratory Objectives



# 3 STUDY OVERVIEW

#### 3.1 Study Design

This Phase 1b/2, multicenter, open-label study was designed to evaluate the efficacy and safety of acalabrutinib in subjects with recurrent GBM who had progressed after 1 or

Acerta Pharma 

Statistical Analysis Plan: ACE-ST-209


2 prior systemic treatment regimens. Subjects meeting the eligibility criteria for the study were assigned 1:1 to one of the following cohorts:

Cohort 1: acalabrutinib 200 mg administered PO BID

Cohort 2: acalabrutinib 400 mg administered PO QD

Under original protocol, an interim analysis was scheduled after the 12 bubject was enrolled in each arm (n=24). If acceptable safety and efficacy (e.g., 2 or more of the 12 subjects [≥ 16.7%] achieve a complete response [CR] or partial response [PR]; additional criteria may be considered by the SAC) are observed in either cohort, the sponsor may choose to expand the study to a total of 72 subjects. The acalabrutinib dosage for the Phase 2 portion of the study will be based on available safety and efficacy data from the Phase 1b cohorts. However, due to the paucity of EIAED-treated subjects, an interim analysis was held after 16 non-EIAED subjects and 1 subject on EIAED were enrolled in the study. The first interim analysis did not raise any safety concerns and showed some response in the 200 mg BID group, while no response in 400 mg QD group. Therefore, the SAC recommended discontinuing Cohort 2 (400 mg QD) and enrolling 7 additional non-EIAED subjects planned for Phase 1b of the study into Cohort 1 (200 mg BID). Under amendment 2 of the protocol, a second interim analysis for safety and efficacy was performed after enrolling an additional 7 subjects, once 15 total subjects enrolled in the 200 mg BID cohort (8 subjects enrolled prior to first interim analysis, and an additional 7 subjects planned to complete Phase 1b).

Under amendment 2 of the protocol, the efficacy criteria for success for phase 1b was as follows: an ORR rate of 3/15 (20%) with a lower bound of a 1-sided 90% exact binomial confidence interval of 7.1% would warrant a recommendation to expand study to phase 2 an enroll additional 28 subjects. Using these criteria, a lower bound of confidence interval of 7.1% would be greater than 5% (ORR estimate for the standard of care CCNU). Based on these criteria, the SAC and the Safety Review Committee did not recommend continuing the study (initiating Phase 2) after reviewing the results of the 2<sup>nd</sup> interim analysis.

Refer to Amendment 2.0 section 3.0 for more details.

#### 3.2 Sample Size

The sample size for the overall study included subjects enrolled in Phase 1b and Phase 2 treated with the same dose regimen. An ORR observed in standard of care for second-line therapies (CCNU) ranged around 5 to 10%. While bevacizumab (Avastin)

Acerta Pharma 

Statistical Analysis Plan: ACE-ST-209


demonstrated an ORR > 20%, considerable toxicities were reported. To reject the null hypothesis of ORR  $\leq$  5% in favor of an alternative hypothesis that the ORR is  $\geq$  20%, 43 subjects will preserve approximately 88% power to detect the difference at a 0.025 significance level by a 1-sided exact test.

However, the initiation of part 2 of the study was dependent on the results of part 1b. The sample size for part 1b was chosen empirically to be 24 subjects. Furthermore, the sample size for subjects treated with acalabrutinib dose of 200mg BID was 15, while 9 subjects were treated with acalabrutinib dose of 400 mg. The sample size and design changes for part 1b are summarized in the table below:

**Table 1 Phase 1b Sample Size Summary** 

| | | Phase 1b | |
|--------------------|-----------|-----------|-------------------------|
| Cohort | | Scheduled | Overall Enrollment |
| Cohort 1: | EIAED* | n = 4 | n = 0 |
| ACP-196 200 mg BID | Non EIAED | n = 8 | n = 15 |
| | | | (7 additional patients) |
| Cohort 2 | EIAED* | n = 4 | n = 1 |
| ACP-196 400 mg QD | Non EIAED | n = 8 | n = 8 |

<sup>\*</sup>EIAEDs are no longer considered the standard of care for patients with glioblastoma.

This SAP includes Phase 1b safety and efficacy analysis that will be performed on the 24 total subjects in Phase 1b comprising the 9 subjects enrolled in the 400 mg QD cohort and the 15 subjects enrolled in the 200 mg BID cohort (8 subjects enrolled prior to first interim analysis, and an additional 7 subjects completing Phase 1b).

Refer to Amendment 2.0 section 5.1 for more details.

#### 4 STUDY ENDPOINTS

### 4.1 Safety Endpoints

The safety of acalabrutinib will be characterized by the type, frequency, severity, timing of onset, duration, and relationship to study drug of any treatment-emergent adverse events (TEAEs) or abnormalities of laboratory tests; study drug-related adverse events (AEs), serious adverse events (SAEs), AEs leading to dose modification, dose delay and discontinuation of study treatment.

Refer to Amendment 2.0 section 5.4.1 for more details.

Acerta Pharma 

Statistical Analysis Plan: ACE-ST-209


#### 4.2 Efficacy Endpoints

Efficacy will be evaluated based on assessments of tumor response and progression using RANO criteria (Wen 2010).

Efficacy endpoints will include:

- Overall response rate (ORR)
- Duration of response (DOR)
- Progression-free survival (PFS)
- 6-month progression-free survival (PFS-6)
- 4-month progression-free survival (PFS-4)
- OS

# 4.3 Exploratory Endpoints

#### 5 HYPOTHESES AND MULTIPLICITY

No hypothesis will be tested and no multiplicity adjustments will be made.

#### 6 ANALYSIS SETS

#### 6.1 Safety Analysis Set

All efficacy and safety analysis will be performed using the safety population, which consists of all subjects who receive any amount of acalabrutinib. The analysis of DOR will only include subjects who have achieved objective response.

# 6.2 Pharmacokinetic/Pharmacodynamic Analyses Set(s)

Pharmacokinetic/Pharmacodynamic evaluable analysis set will be defined by PK and PD group.

#### 7 SUBGROUP ANALYSIS

NA.

#### 8 FINAL ANALYSIS AND CLINICAL STUDY REPORT

Planned final analysis will be conducted once last subject exits study, or sponsor decides to close the study, whichever occurs earlier.

#### 9 MISSING VALUES

No imputation of values for missing data will be performed except for missing or partial

Acerta Pharma 

Statistical Analysis Plan: ACE-ST-209


dates according to prespecified, conservative imputation rules. The details of imputation rules for partial or missing dates are listed in Appendix 12.2.

#### 10 STATISTICAL METHODS OF ANALYSIS

#### 10.1 General Principles

Descriptive statistics [including sample size, group means, standard deviations, medians, minimum and maximum for continuous variables and sample size, frequency, proportions and confidence intervals (CIs) for discrete variables] will be used to summarize will be used to summarize data as appropriate.

Calculation of time to event or duration of event endpoints will be based on the study day of the event or censoring date rather than visit number or visit label. Missing efficacy or safety data will not be imputed unless otherwise specified.

The following rules will be used for the days to months/years conversion:

- 1 month= 30.4375 days;
- 1 year= 365.25 days.

All summaries will be presented by treatment cohort.

#### 10.2 Subject Accountability

The number of subjects enrolled by site, country and region (US and ex-US) will be presented. Subject disposition will be summarized for all enrolled subjects including the following information:

- Proportion of subjects who received study drug
- Proportion of subjects with study drug discontinuation and primary reason for study drug discontinuation
- Proportion of subjects discontinuing study and reasons for study discontinuation
- Time on study

#### 10.3 Important Protocol Deviations

Important Protocol Deviations (IPDs) categories are defined and managed by the study team during the IPD reviews throughout the study before database lock. The final IPD list for each study is used to produce the summary of IPDs table and the listing of subjects with IPDs, respectively.

#### 10.4 Demographic and Baseline Characteristics

Summaries of demographic characteristics will be presented for age, age category (< 65, ≥ 65), gender, race, ethnicity, and geographic region.

Acerta Pharma 

Baseline characteristics will be presented for Eastern Cooperative Oncology Group (ECOG) performance status, disease stage, tumor grade, number of prior anticancer therapies.

#### 10.5 Treatment and Medications

#### 10.5.1 Prior Anticancer Therapies

Summary statistics will be presented for prior anticancer regimens (might include multiple therapies) and prior cancer-related surgery. The number of lines and type of prior therapy will be summarized.

#### 10.5.2 Concomitant Medications

Concomitant medications will be coded and tabulated according to the World Health Organization (WHO) Drug Dictionary (WHODRUG).

#### 10.5.3 Exposure to Investigational Product

The number of subjects who received at least one dose of acalabrutinib, duration of exposure, average daily dose, and relative dose intensity will be summarized by treatment cohort.

Exposure parameters are defined in more detail in Appendix 12.1.

#### 10.6 Safety Analyses

All safety analysis will be performed using the safety analysis set.

#### 10.6.1 Adverse Events

The Medical Dictionary for Regulatory Activities (MedDRA v20.1 or later) will be used to code all AEs to a system organ class and a preferred term. The severity of the AE will be assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. Study drug-related AEs are those assessed by investigator as related.

All AE tables will be summarized by treatment cohort.

TEAEs are defined as those events that occur or worsen on or after the first dose of study drug(acalabrutinib), through the treatment phase, and within 30 days following the last dose of acalabrutinib.

TEAEs will be summarized by system organ class (SOC) and preferred terms (PTs) as well as preferred terms only in descending order of frequency, by CTCAE severity grade.

Acerta Pharma 

Statistical Analysis Plan: ACE-ST-209


Drug-related TEAEs, treatment-emergent serious adverse events (TESAEs), TEAEs leading to study drug discontinuation or dose modifications or dose delay will be summarized by PTs in descending order of frequency and by CTCAE severity grade.

Death information is reported in the study exit case report form (CRF) and death information CRF for all deaths. Incidences of deaths are to be reported, along with the primary cause of death.

#### 10.6.2 Events of Clinical Interest

Broader categories of Events of Clinical Interest (ECI) identified for acalabrutinib will be summarized. The definitions of these categories for safety analysis are part of Appendix 12.5.1 and Appendix 12.5.2.

#### 10.6.3 Laboratory Test Results

Laboratory data up to 30 days after last dose or the safety follow-up visit date, whichever is later, will be reported in International System of Units (SI) units. Applicable laboratory results will be graded according to CTCAE Version 4.03. For each laboratory parameter, the baseline laboratory value/grade is defined as the last laboratory value/grade collected on or prior to the date of the first dose of study drug. Treatment-emergent laboratory abnormalities for selected parameters will be summarized.

## 10.6.4 Vital Signs

Body temperature, heart rate (beats/min), systolic blood pressure (mmHg), diastolic blood pressure (mmHg), respiratory rate (breaths/min), and weight will be collected for each study as scheduled in Amendment 2 Appendix 1. Schedule of Assessments. For each parameter, summary statistics (mean, standard deviation, median, and range) will be produced for baseline, maximum, and minimum value.

#### 10.6.5 ECOG Performance Status

ECOG performance status scores will be summarized for each treatment cohort using shift table. The shifts in scores from baseline to worst ECOG score on treatment will be summarized.

#### 10.7 Efficacy Analyses

All efficacy analysis will be performed using the safety analysis set. The analysis of DOR will only include subjects who have achieved objective response.

Statistical Analysis Plan: ACE-ST-209


# 10.7.1 Best Overall Response, Disease Control Rate and Overall Response Rate per RANO criteria

Measurable disease (bidimensional) as defined by the RANO criteria. RANO criteria (Wen 2010) will be followed for selection of measurable and non-measurable lesions and about the number of lesions to be assessed, as well as for the assessments of response and progression.

Disease Control Rate (DCR) is defined as the proportion of subjects who achieve a best response of SD, PR or CR at any point of the study.

Overall response Rate (ORR) is defined as the proportion of subjects who achieve a best response of PR or CR at any point of the study.

The primary analysis of DCR and ORR will be conducted using safety analysis set. DCR and ORR will be calculated with the corresponding exact binomial 2-sided 95% CI and 1-sided 90% CI (or 2-sided 80% CI) for treatment cohort.

# 10.7.2 Duration of Response per RANO criteria

The DOR is defined as the interval from the first documentation of response to the earlier of the first documentation of definitive disease progression or death from any cause. The DOR will be summarized appropriately for subjects in safety analysis set who achieved response (CR or PR) at any point of the study. Kaplan-Meier methods will be used to estimate event-free curves and corresponding quantiles (including the median).

Data from surviving, non-progressing subjects will be censored at the date of the last adequate disease assessment that is on or before the start date of the new antitumor therapy. Data from subjects who have disease progression or die after more than one missed visit will be censored at the last visit date before the missing assessments which lack objective disease assessment. The details of definition of progression events and censoring rules are the same as for PFS endpoint and are listed in <u>Appendix 12.3</u>

# 10.7.3 Progression-free Survival Per RANO criteria

Progression-free survival is defined as the interval from the start of therapy to the earlier of the first documentation of objective disease progression or death from any cause,

Statistical Analysis Plan: ACE-ST-209


whichever occurs first. Kaplan-Meier (K-M) methods will be used to estimate the event-free curves and corresponding quantiles (including the median).

Data from surviving, non-progressing subjects will be censored at the date of the last adequate disease assessment that is on or before the start date of the new antitumor therapy. Data from subjects who have disease progression or die after more than one missed visit will be censored at the last visit date prior to the missing assessments which lack objective disease assessment. The details of definition of progression events and censoring rules are listed in Appendix 12.3.

In the primary analysis using safety analysis set, study treatment end date will be used as the date of progression for subjects who discontinued study treatment due to disease progression or death prior to 1<sup>st</sup> radiographic assessment. Data for subjects who discontinued study treatment prior to 1<sup>st</sup> radiographic assessment due to reasons other than disease progression or death will be censored at their study treatment start date.

# 6-month Progression-free Survival (PFS-6) Rates and 4-month Progression-free Survival (PFS-4) Rates

PFS-6 rate is defined as the K-M estimate of subjects alive and without documented disease progression at 6 months. The K-M method will be used to estimate the PFS-6 rate and corresponding exact 2-sided 95% CIs. The same method applies to the PFS-4 rate.

#### 10.7.4 Overall Survival

Overall survival is defined as the time from date of enrollment until date of death due to any cause. Subjects who are known to be alive or whose survival status is unknown will be censored at the date last known to be alive. Subjects who lost to follow-up for survival immediately after randomization will be censored at first dose date.

OS will be summarized for safety analysis set. The analysis methods for OS will be similar to those described for progression-free survival. Censoring rules are defined in more detail in Appendix 12.4.

Acerta Pharma 

Statistical Analysis Plan: ACE-ST-209


# 10.7.5 Pharmacokinetic, Pharmacodynamic and Biomarker Analyses

Additional pharmacodynamic, pharmacokinetic and biomarker analyses may be performed, as deemed appropriate. A separate analysis plan for these analyses will be developed by PK/PD group at Acerta.

Acerta Pharma 

Statistical Analysis Plan: *ACE-ST-209* Version *1.0* dated:07 *April 2018* 

#### 11 LITERATURE CITATIONS / REFERENCES

 Guidance for Industry. Clinical Trail Endpoints for the Approval of Cancer Drugs and Biologics. FDA. May 2007. <a href="http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/ucm071590.pdf">http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/ucm071590.pdf</a>

- Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0, USDHHS, NIH, NCI; publish date May 28, 2009 (v4.03: June 14, 2010).
- Patrick Y. Wen, David R. Macdonald, David A. Reardon, et al. Updated Response Assessment Criteria for High-Grade Gliomas: Response Assessment in Neuro-Oncology Working Group. J Clin Oncol 28:1963-1972

Acerta Pharma 

Statistical Analysis Plan: ACE-ST-209


#### 12 APPENDICES

#### 12.1 Definitions

## Study Day

The study day will be calculated in reference to the first dose date of study drug. Study Day 1 is defined as the first dose date of study drug. For assessments that occur on or after the first dose date of study drug, study day is defined as (date of assessment – first dose date of study drug + 1). For assessments that occur prior to the first dose date of study drug, study day is defined as (date of assessment – first dose date of study drug). There is no Study Day 0.

#### **Duration of Exposure**

The duration of exposure to acalabratinib will be calculated in months as (last dose date - first dose date + 1) / 30.4375. The gaps in treatment will be included. The duration of exposure in days will be used for planned dose calculation.

#### **Total Dose**

Total dose received is a sum of all actual doses taken through the treatment duration and will be presented in grams. For scheduled drug administration visits that are skipped the actual dose will be 0.

#### Average Daily Dose

Average daily dose is total dose divided by duration of exposure in days.

#### Relative Dose Intensity

Relative dose intensity is the ratio of total dose to the protocol-specified total dose through the duration of exposure.

Acerta Pharma 

Statistical Analysis Plan: ACE-ST-209


# 12.2 Imputation rules for partial or missing dates

Imputation of partial dates will be made for AE onset and stop dates, start and end dates of concomitant medication, start date of subsequent anticancer therapy, date of initial diagnosis and death date. If dates are completely missing, no imputation will be made. For any partial date with missing year, no imputation will be made.

The general rule for imputation is:

- If only day is missing, then the 15<sup>th</sup> of the month will be used.
- If only year is present, then June 30<sup>th</sup> will be used.

If such imputation date for initial diagnosis is on or after date of first dose, then date of first dose – 1 will be used. If such imputed date for subsequent anticancer therapies is before date of last dose, then date of last dose + 1 will be used.

If the imputed date is for an AE start date and is in the same year and month as but before the first dose date, then the first dose date will be used, or if the imputed AE start date is after the AE end date, then the AE end date will be used. If the imputed date is for an AE start date and is in the same year and month as but after the last dose date + 30 days, then the last dose date + 30 days will be used.

If the imputed date is for an AE end date and is after the death date, then the death date will be used, or if the imputed AE end date is before the AE start date, then the AE start date will be used.

Every effort will be made to obtain complete dates for deaths. If both month and day are missing for death date or a death date is totally missing, do not impute and censor the subject survival time. If death year and month are available but day is missing, the following algorithm will be used:

- If mmyyyy for last contact date = mmyyyy for death date, set death date to the day after the last contact date.
- If mmyyyy for last contact date < mmyyyy for death date, set death date to the first day of the death month.
- If mmyyyy for last contact date > mmyyyy for death date, data error and do not impute.

Acerta Pharma 

Statistical Analysis Plan: ACE-ST-209


# 12.3 PFS events and censoring rules

Here PFS is the primary analysis that only includes well-documented and verified progression events.

Same rules are used for DOR identify progression or censoring date.

| Situation | PFS | |
|---|---|---|
| | Date of Progression or Censoring | Outcome |
| Progression documented on<br>scheduled visit | Date of scheduled visit | Progression |
| Progression documented between scheduled visits | Date of unscheduled visit | Progression |
| Treatment discontinuation for undocumented progression | Date of last visit with adequate assessment | Censor |
| Death before first PD assessment | Date of death | Progression |
| Death between adequate assessment visits | Date of death | Progression |
| Death or progression after only one missed visit | Date of death | Progression |
| Death or progression after 2 or more missed visits | Date of last visit with adequate assessment | Censor |
| Death or progression after 2 or<br>more missed visits and only<br>baseline tumor assessment<br>available | Date of 1st dose of study drug | Censor |
| No baseline tumor assessments | Date of 1st dose of study drug | Censor |
| Baseline tumor assessments<br>only and no evidence of<br>documented PD, treatment<br>discontinuation due to PD or<br>death within no more than one<br>missed visit | Date of 1st dose of study drug | Censor |
| No progression | Date of last visit with adequate assessment | Censor |
| Treatment discontinuation for toxicity or other reason | Date of last visit with adequate assessment | Censor |
| New anticancer treatment started | Date of last visit with adequate assessment | Censor |

Acerta Pharma 

Statistical Analysis Plan: *ACE-ST-209* Version *1.0* dated:07 *April 2018* 

#### 12.4 Overall survival censoring rules

| Situation | Date Death or Censoring | Outcome |
|---|---|---|
| Death at any timepoint | Date of death | Death |
| Lost to follow-up immediately after 1st dose of study drug | Date of 1st dose study drug | Censored |
| Not known to have died at or after the analysis cutoff date | The date last known alive before data analysis cutoff | Censored |
| Known to have died after the analysis cutoff date | Date of data analysis cutoff | Censored |

Acerta Pharma 

Statistical Analysis Plan: *ACE-ST-209* Version *1.0* dated:07 *April 2018* 

#### 12.5.1 Events Of Clinical Interest

The Events of Clinical Interest (ECIs) have been identified based on preclinical findings, emerging data from clinical studies relating to acalabrutinib, and pharmacological effects of approved BTK inhibitor. The AEs selected for dedicated analysis were evaluated using Standardized MedDRA Queries (SMQs), where available, by SOC, or by Sponsor-defined baskets of MedDRA Adverse Event Grouped Terms.

| Category name | Sub-category name | Definition |
|---|---|---|
| Cardiac events | | SOC Cardiac disorders |
| | Atrial fibrillation | PT Atrial fibrillation |
| | | PT Atrial flutter |
| Cytopenias – Anemia | | SMQ Haematopoietic erythropenia [narrow + broad] |
| Cytopenias – Leukopenia | | SMQ Haematopoietic leukopenia [narrow + broad] |
| | Neutropenia | PT Febrile Neutropenia |
| | | PT Neutropenia |
| | | PT Neutropenic infection |
| | | PT Neutropenic sepsis |
| | | PT Neutrophil count decreased |
| | | PT Neutrophil percentage decreased |
| | Other Leukopenia | SMQ Haematopoietic leukopenia [narrow + broad]<br>excluding PTs for neutropenia above |
| Cytopenias -<br>Thrombocytopenia | | SMQ Haematopoietic thrombocytopenia [narrow + broad] |
| Hemorrhage | | SMQ Haemorrhage terms (excl laboratory terms) |
| | Major hemorrhage | As per Acerta definition in Appendix 12.5.2 below |
| Hepatic Events | | <ul> <li>SMQ [narrow] Hepatic failure, fibrosis and cirrhosis<br/>and other liver damage-related conditions</li> </ul> |
| | | SMQ [narrow] Liver related investigations signs |
| | | SMQ [narrow] Hepatitis, non-infectious |
| Hypertension | | SMQ Hypertension [narrow] |
| Infections | | SOC Infections and infestations |
| Interstitial lung disease/Pneumonitis | | SMQ [narrow] Interstitial lung disease |
| Second primary<br>malignancies | | SMQ Malignant or unspecified tumours and SMQ Myelodysplastic syndrome [narrow] |
| | Second primary<br>malignancies<br>(excluding skin) | SMQ Malignant or unspecified tumours and SMQ<br>Myelodysplastic syndrome [narrow], excluding skin<br>(i.e. exclude SMQ Skin neoplasms, malignant and<br>unspecified) |
| Tumor lysis syndrome | | PT Tumour lysis syndrome |

MedDRA version 20.1

Acerta Pharma 

<sup>&#</sup>x27;No additional criteria' means only SAE, AE leading to study drug discontinuation, and deaths within specified window will be selected for narratives.

<sup>&#</sup>x27;Any' means any subject with a PT in the category will be selected for narratives.

Statistical Analysis Plan: ACE-ST-209


#### 12.5.2 Major Hemorrhage

Major hemorrhage is defined as any hemorrhagic event that is serious, or Grade  $\geq$  3 in severity, or that is a central nervous system (CNS) hemorrhage (any severity grade).

# Search Strategy:

- Use standardized MedDRA v20.1 Query:
  - o Haemorrhage terms (excl laboratory terms) (SMQ) [20000039]
- II. Identify Major Events that are a subset of the Haemorrhage SMQ:
  - o Grade ≥ 3 AE
  - o Any SAE
  - All Grades of CNS hemorrhage

CNS hemorrhage Preferred Terms (MedDRA v20.1):

| CNS hemorriage Freierred Terms (MedDRA V20.1). | |
|---|---|
| Acute haemorrhagic leukoencephalitis | Haemorrhagic transformation stroke |
| Basal ganglia haematoma | Intracerebral haematoma evacuation |
| Basal ganglia haemorrhage | Intracranial haematoma |
| Basilar artery perforation | Intracranial tumour haemorrhage |
| Brain contusion | Intraventricular haemorrhage |
| Brain stem haematoma | Intraventricular haemorrhage neonatal |
| Brain stem haemorrhage | Meningorrhagia |
| Brain stem microhaemorrhage | Ocular retrobulbar haemorrhage |
| Central nervous system haemorrhage | Optic disc haemorrhage |
| Cerebellar haematoma | Optic nerve sheath haemorrhage |
| Cerebellar haemorrhage | Periventricular haemorrhage neonatal |
| Cerebellar microhaemorrhage | Pituitary haemorrhage |
| Cerebral aneurysm perforation | Putamen haemorrhage |
| Cerebral aneurysm ruptured syphilitic | Ruptured cerebral aneurysm |
| Cerebral arteriovenous malformation haemorrhagic | Spinal cord haematoma |
| Cerebral artery perforation | Spinal cord haemorrhage |
| Cerebral haematoma | Spinal epidural haematoma |
| Cerebral haemorrhage | Spinal epidural haemorrhage |
| Cerebral haemorrhage foetal | Spinal subarachnoid haemorrhage |
| Cerebral haemorrhage neonatal | Spinal subdural haematoma |
| Cerebral microhaemorrhage | Spinal subdural haemorrhage |
| Encephalitis haemorrhagic | Subarachnoid haematoma |
| Epidural haemorrhage | Subarachnoid haemorrhage |
| Extradural haematoma | Subarachnoid haemorrhage neonatal |
| Haemorrhage intracranial | Subdural haematoma |
| Haemorrhagic cerebral infarction | Subdural haematoma evacuation |
| Haemorrhagic stroke | Subdural haemorrhage |
| Subdural haematoma evacuation | Subgaleal haematoma |
| Subdural haemorrhage | Thalamus haemorrhage |
| Subdural haemorrhage neonatal | Traumatic intracranial haemorrhage |

Acerta Pharma 